CLINICAL TRIAL: NCT06207214
Title: Acceptance and Commitment Therapy for University Students: A Single Case Experimental Study of the Self-help Book "The Unbreakable Student"
Brief Title: Evaluating an ACT Self-help Book for University Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff University (Other)
Responsible Party: Principal Investigator, Victoria Phillips, Principal Investigator (Trainee Clinical Psychologist), Cardiff University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ACTSelfHelpBookStudents2023
Record Dates: First submitted 2023-11-22; First posted 2024-01-16 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Well-Being, Psychological
Keywords: Acceptance and Commitment Therapy; Self-help; University students; Single Case Design
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-help book for University Students (Experimental): The Unbreakable Student: 6 Rules for Staying Sane at University by Dr Nic Hooper.
  Interventions: Other: Self-help book for university students.

INTERVENTIONS:
Other: Self-help book for university students. — The intervention being tested, is a self-help book for university students based on Acceptance and Commitment Therapy. The book was published in 2021 and is called "The Unbreakable Student: 6 Rules for Staying Sane at University". The book is by Dr Nic Hooper.
  The self-help book will be posted in paper form to all participants. There are 8 chapters in the book and participants will be given eight weeks to read the book at home (with a suggestion of reading one chapter per week).

SUMMARY:
Background to the project:

More and more university students are reporting poor mental health, which has resulted in long waiting lists for student support services. Given this context, self-help solutions, (which means giving students ideas in books/apps/websites that they can try in their own time to help with their problems), are becoming more important.

Rationale for the project:

There are many self-help resources for students but not many of them are well-researched. This research project will test a self-help book called "The Unbreakable Student: 6 Rules for Staying Sane at University".

Methodology:

A small group of students (approximately 12) will complete questionnaires at three time points (prior to reading the book, whilst reading the book and after reading the book). They will also answer four questions sent via text message, every three days throughout the study. These will relate to a particular aspect of university life which they have identified as stressful. They will also be interviewed afterwards, to give information about their experiences of reading the book and use of the end of chapter tasks etc.

Purpose:

The purpose is to find out if the book is helpful for students and, if so, which parts were the most helpful.

Hypotheses:

The book will help students to be less bothered by difficult thoughts, such that they might find them less interfering and may feel more engaged in meaningful activities.

The book will also improve student wellbeing.

DETAILED DESCRIPTION:
Aims:

The proposed research aims to assess whether reading "The Unbreakable Student: 6 Rules for Staying Sane at University" leads to any changes in idiosyncratic student outcomes, measures of student wellbeing and ACT based processes amongst a student population. It also aims to explore when in the intervention, any differences occur, to determine which content leads to the most change for students and therefore which change mechanisms should be targeted or prioritised in future student interventions.

Hypotheses:

It is hypothesised that reading an ACT based self-help book will change the way students relate to their experiences and thoughts about university stress. It is hypothesised that there will not be a significant change in how regularly students think about their source of stress. It is hypothesised that there may be a reduction in how interfering students rate their thoughts about a stressful topic and an increase in how they rate their engagement in meaningful activities, in spite of the stressors they face. These hypotheses will be tested via the use of idiosyncratic target variables.

It also hypothesised that there will be an increase in overall student wellbeing and ACT related processes, as measured by nomothetic measures.

Methodology and outcome measures:

The overall study design will be a Single Case Experimental Design (SCED) approach.

There will be an initial baseline phase, where participants will each complete idiosyncratic measures every three days. Participants will be randomly allocated to a baseline phase of either 2, 3 or 4 weeks. The idiosyncratic measures will use a Likert scale format and will assess frequency of thoughts, level of interference of thoughts and ability to engage in meaningful activities despite the thoughts. These will all be personalised to individual participants, as per their individual target problem/source of stress, which they will have identified during a screening phase. These will act as dependent variables. The baseline phase will be monitored for stability. After this, the independent variable will be introduced, and participants begin reading "The Unbreakable Student: 6 Rules for Staying Sane at University". Participants will be given 8 weeks to read the book (which has 8 chapters) and participants will be suggested to read 1 chapter a week. Participants continue completing their idiosyncratic measures, every three days, throughout the intervention phase.

Participants will also complete nomothetic measures. These will be the Warwick-Edinburgh Mental Well-being Scale - WEMWBS (to assess student wellbeing) and the COMPrehensive assessment of Acceptance and Commitment Therapy processes - the CompACT measure (to assess ACT processes). These will be completed pre-intervention, mid-intervention and post-intervention. Demographic data will also be collected (e.g. gender, age, course subject and year of study).

Post-intervention there will be exit interviews; to discuss the findings, assess any external confounding events and explore student participation in the end of chapter tasks. These would use a semi-structured interview schedule. They would be recorded and transcribed via Teams and would be analysed using (descriptive) thematic analysis.

Participants:

The aim will be to recruit between six and 12 participants. In single case designs, students act as their own controls, meaning the intervention can be tested using a small sample and evaluated more robustly than in an uncontrolled case study. This avoids needing a large student to read an entire book (due to issues with student research participation). Participants will predominantly be recruited via social media.

Screening:

Participants will complete an online screening questionnaire, to assess eligibility for the study. The screening questionnaire will:

* Check they are registered as a Cardiff University student.
* Check they have no links with the author of the book.
* Check anything that would impact their ability to read a book (e.g. language/disability) and any adjustments required.
* Identify an area of stress that the student has, in relation to their university experience.
* Check they have not previously read the book.
* Check they are not taking part in any other research studies or interventions that could confound the results.
* Use the Clinical Outcomes in Routine Evaluation 10 (CORE-10) measure to check there is no significant clinical risk.

Intervention:

The intervention being tested, is a self-help book for university students based on Acceptance and Commitment Therapy. The book was published in 2021 and is called "The Unbreakable Student: 6 Rules for Staying Sane at University". The book is by Dr Nic Hooper.

Data analysis:

The hypotheses will be tested using visual inspection, as per usual data evaluation in SCED and also by statistical methods (such as Tau/PAND). These will be used to analyse the idiosyncratic data. Furthermore, clinically significant change and reliable change will be measured, and will used to analyse data from the standardised/nomothetic psychometric measures. The interviews will be analysed using thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Registered as a current Cardiff University student.
* Proficient in English.
* Have an adequate reading level.
* Identify as experiencing a non-clinical, university or study related difficulty. Examples include: Exam/presentation nerves, feelings of loneliness/stress/anxiety/low mood, binge drinking, procrastination, feelings of burnout, academic/course worries, unhealthy lifestyle choices.

Exclusion Criteria:

* Must not be a Cardiff University psychology student, due to potential social desirability bias, associated with being from the same school as the book author.
* Must not have read "The Unbreakable Student: 6 Rules for Staying Sane at University".
* Must not be in concurrent research studies/receiving concurrent psychological support, including psychoeducational, therapeutic or self-help interventions. This is to ensure valid conclusions can be drawn about the impact of the book.
* Must not present with heightened risk during recruitment, as screened for by the CORE-10. This will be defined as a score within the moderate-severe/severe range (which is a score of 20 or higher) and/or indication of suicidal intent as indicated on the risk item. This is to ensure participant safety, whilst also ensuring a sample that reflects current levels of student distress. Any students not eligible due to risk will be signposted to services such as student support or their General Practitioner (GP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-02-24 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Frequency of thoughts about idiosyncratic stressor. | Participants will complete this measure every 3 days, for the duration of their baseline phase (randomly allocated) and for the duration of the intervention phase (8 weeks).
  Participants will be asked to rate how often they have had thoughts about their idiosyncratic stressor, on a scale of 0-10 (0 = not very often at all, 10 = all the time).
Impact of thoughts about idiosyncratic stressor. | Participants will complete this measure every 3 days, for the duration of their baseline phase (randomly allocated) and for the duration of the intervention phase (8 weeks).
  Participants will be asked to rate how interfering their thoughts about their idiosyncratic stressor have been, on a scale of 0-10 (0 = not interfering at all, 10 = very interfering).
Engagement in meaningful activities. | Participants will complete this measure every 3 days, for the duration of their baseline phase (randomly allocated) and for the duration of the intervention phase (8 weeks).
  Participants will be asked to rate how engaged they feel in meaningful activities, in spite of any thoughts about their idiosyncratic stressor, on a scale of 0-10 (0 = not very engaged, 10 = fully engaged).

SECONDARY OUTCOMES:
Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) | Baseline, mid-intervention (week 4 of the book reading phase) and follow-up (1 week after completing the book reading phase).
  Measure of overall wellbeing. Minimum score is 14 and maximum score is 70. A higher score indicates better wellbeing outcomes.
Comprehensive assessment of Acceptance and Commitment Therapy processes (CompACT) | Baseline, mid-intervention (week 4 of the book reading phase) and follow-up (1 week after completing the book reading phase).
  Measure of psychological flexibility. For this measure, participants rate items on a 7-point Likert scale (which goes from 0 meaning strongly disagree, to 6, meaning strongly agree), with some items being reversed scored.
  Scores are then calculated for each of the subscales (openness to experience, behavioural awareness, valued action) and a total score is completed by adding these together.
  The minimum score is 0 and the maximum score is 138. A higher score on this measure, represents greater psychological flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Phillips, Principal Investigator — Cardiff University
Locations (1):
- Based at Cardiff University (study to be completed remotely), Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All data will be retained in line with Cardiff University's Records Retention Schedule.
  The research team also aim to publish this project in a relevant journal, upon completion of the write-up. Any data made available as part of this publication process, will be fully anonymised.
Supporting Information: Study Protocol, SAP
Time Frame: Any anonymised data which is included as part of the final report, will be made available from the point of publication and will be in the public domain indefinitely. All other data stored by Cardiff University, will be managed in line with the Records Retention Schedule.

REFERENCES:
- [Background] Braun, V., & Clarke, V. (2006). Using thematic analysis in psychology. Qualitative research in psychology, 3(2), 77-101. https://doi.org/10.1191/1478088706qp063oa
- [Background] Morley S. (2017). Single case methods in clinical psychology: A practical guide. Routledge.
- [Background] Kazdin AE. Single-case experimental designs. Evaluating interventions in research and clinical practice. Behav Res Ther. 2019 Jun;117:3-17. doi: 10.1016/j.brat.2018.11.015. Epub 2018 Dec 2. PMID 30527785
- [Background] Stewart-Brown S, Evans J, Patterson J, Petersen S, Doll H, Balding J, Regis D. The health of students in institutes of higher education: an important and neglected public health problem? J Public Health Med. 2000 Dec;22(4):492-9. doi: 10.1093/pubmed/22.4.492. PMID 11192277
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127
- [Background] Morley, S., Dowzer, C.N. (2014) Manual for the Leeds Reliable Change Indicator: Simple excel applications for the analysis of individual patient and group data. University of Leeds, Leeds, UK.